CLINICAL TRIAL: NCT07294937
Title: Study Protocol: 10-Year Follow-Up of Patients Screened for Cardiovascular Risk by the "All With Heart" Association - Development of a Morocco-Specific Risk Score
Status: Recruiting | Type: Observational
Sponsor: Moroccan Society of Cardiology (Other)
Collaborators: F&C Clinical Trials (Unknown)
Responsible Party: Sponsor
Other Study IDs: 126/24
Record Dates: First submitted 2025-12-02; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases (CVD)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants screened for cardiovascular risk (TAC cohort): Participants aged 40 years and older who were screened for cardiovascular risk between 2010 and 2012 by the "All with heart" Association in the Greater Casablanca region. This cohort is being followed 10 years after the initial screening to assess cardiovascular outcomes (death, myocardial infarction, stroke) and to develop a Morocco-specific cardiovascular risk score. No intervention is applied; the study is purely observational.

SUMMARY:
Cardiovascular diseases (CVDs) are the leading cause of death worldwide, and their prevalence is steadily increasing in Morocco. Between 2010 and 2012, the "All with heart" Association conducted a large-scale cardiovascular screening campaign in the Greater Casablanca region, involving more than 10,000 adults aged over 40 years. This 10-year follow-up study aims to evaluate long-term cardiovascular outcomes and to develop a Morocco-specific cardiovascular risk score. Follow-up data will be collected through phone calls, WhatsApp, or SMS with participants or their families to document cardiovascular deaths, myocardial infarctions, and strokes. Statistical analyses, including survival analysis and multivariate logistic regression, will be used to identify significant risk factors and to construct a predictive risk model tailored to the Moroccan population. The study received a favorable opinion from the Rabat Ethics Committee. Written informed consent will be obtained from all participants or their families prior to data collection. The findings are expected to enhance understanding of cardiovascular risk evolution in Morocco and to provide a validated, population-specific risk score to support prevention and patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years or older at the time of the initial screening (2010-2012).
* Individuals who participated in the cardiovascular risk screening campaign conducted by the "All with heart" Association between 2010 and 2012 in the Greater Casablanca region.
* Moroccan nationality.
* Participants or family members who provide written informed consent for participation in the 10-year follow-up study.

Exclusion Criteria:

* Individuals who refuse to participate in the follow-up study.
* Participants who have moved and cannot be reached by phone, WhatsApp, or SMS.
* Participants who died from non-cardiovascular causes.
* Non-Moroccan participants.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 40 years and older who were screened for cardiovascular risk between 2010 and 2012 by the "All with heart" Association in the Greater Casablanca region, Morocco. Approximately 10,000 individuals participated in the original screening campaign, which collected data on anthropometric, biological, and lifestyle risk factors.
  For the 10-year follow-up, all eligible Moroccan participants from the initial screening will be contacted by phone, WhatsApp, or SMS to collect updated information on cardiovascular events, hospitalizations, and mortality. This population represents a community-based cohort reflecting the general adult population at risk of cardiovascular disease in Morocco.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Cardiovascular Events (MACE) | 10 years after initial screening (2010-2012)
  Occurrence of major cardiovascular events (myocardial infarction, stroke, or cardiovascular death) among participants screened for cardiovascular risk between 2010 and 2012 by the "All with heart" Association. Events will be identified during the 10-year follow-up period through participant or family contact (phone, WhatsApp, or SMS) and verified through available medical records when possible.
Development and Validation of a Morocco-Specific Cardiovascular Risk Score | Baseline (2010-2012) and 10-year follow-up (2022)
  Development and internal validation of the Morocco-Specific Cardiovascular Risk Score, a composite risk prediction score estimating the 10-year probability of major cardiovascular events including myocardial infarction, stroke, or cardiovascular death. The score will be derived from baseline cardiovascular risk factors collected during the initial screening and weighted using multivariable regression models based on outcomes observed during the 10-year follow-up. The score will be expressed on a scale ranging from 0 to 100, where higher scores indicate a higher cardiovascular risk and therefore a worse outcome. Model performance will be assessed using discrimination and calibration measures, including the area under the receiver operating characteristic curve and calibration analyses.

SECONDARY OUTCOMES:
Incidence of Minor Cardiovascular Events | 10 years after initial screening (2010-2012)
  Occurrence of minor cardiovascular events, including stable or unstable angina, among participants screened between 2010 and 2012. Events will be collected through participant or family interviews and verified with medical records when available.

OTHER OUTCOMES:
Number of Hospitalizations Related to Cardiovascular Diseases | 10 years after initial screening (2010-2012)
  Total number of hospitalizations due to cardiovascular causes (acute coronary syndrome, heart failure, arrhythmia, or cardiac surgery) during the 10-year follow-up period.
Change in Cardiovascular Risk Factors Over Time | 10 years after initial screening (2010-2012)
  Change in major cardiovascular risk factors (body mass index, blood pressure, total cholesterol, triglycerides, HDL, blood glucose, smoking status, and physical activity) between the initial screening and the 10-year follow-up.
Quality of Life Assessment | 10 years after initial screening (2010-2012)
  Evaluation of participants' quality of life using a standardized questionnaire (EQ-5D). The assessment will explore mobility, self-care, usual activities, pain/discomfort, and anxiety/depression dimensions.

CONTACTS AND LOCATIONS:
Locations (2):
- Morocco (2):
  - Moroccan Society of Cardiology, Casablanca
  - Cardiology Centre, Mohammed V Military Hospital, Rabat, Morocco, Rabat

IPD SHARING:
Plan to Share IPD: No
The sharing of individual participant data (IPD) is not authorized by the Ethics Committee of Rabat.
  According to the committee's decision, data collected in this study are strictly confidential and may only be used by the research team for the purposes defined in the approved protocol. All collected data will remain stored securely and will not be shared with other researchers or institutions to ensure compliance with national data protection regulations and the ethical approval obtained for this study.